CLINICAL TRIAL: NCT06526013
Title: Cholesterol Self-testing in Patients Post Acute Coronary Syndrome
Acronym: C-Check
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BGAAF-2593
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Acute Coronary Syndrome; Prevention; LDL Hyperlipoproteinemia; Therapeutic Adherence
Keywords: Acute Coronary Syndrome; Dyslipidemia; Statin; Lipid lowering therapy; Cardiovascular disease
MeSH Terms: conditions — Acute Coronary Syndrome; Treatment Adherence and Compliance; Dyslipidemias; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: After randomization into the intervention arm versus control, patients in the intervention group will receive a device for self-measurement and will be trained in its use. Subsequently, these patients will independently measure their cholesterol levels monthly using capillary blood tests and report the results to the study physicians, who will then adjust the therapy accordingly. The control group will attend scheduled visits at months 6 and 12, where medication adjustments can be made, as has been done in the outpatient clinic up to now
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Usual care according to current procedure (in patients with post acute coronary syndrome) regarding LDL target level adjustment
- Cholesterol self-measurement (Experimental): Training patients for self-monitoring of cholesterol, with independent monthly measurements and reporting of results to the study team, followed by prompt therapy adjustments
  Interventions: Other: Cholesterol self-measurement

INTERVENTIONS:
Other: Cholesterol self-measurement — Patients will be trained to use a device to self-measurement of cholesterol-values monthly. After the measurement they will report their results to study team for ajusting the therapy.
  Arms: Cholesterol self-measurement

SUMMARY:
The pharmacological reduction of LDL-C lowers cardiovascular risk and is therefore a priority in cardiovascular secondary prevention. The achievement of LDL-C target levels in Germany, Europe, and worldwide is inadequate, despite a wide array of lipid-lowering medications. Only a small proportion of post-myocardial infarction patients reach their LDL-C target range within a year. There is a significant need for new strategies to improve LDL-C target achievement and thereby reduce the occurrence of secondary cardiovascular events.

The aim of the study is to establish a basis for improving prevention by achieving the target LDL level effectively and quickly in patients with high and very high cardiovascular risk profiles.

DETAILED DESCRIPTION:
In this randomized study, the investigators aim to investigate whether additional self-monitoring of cholesterol values by patients leads to more effective LDL reduction and quicker achievement of the target LDL range versus usual care.

This study systematically and prospectively examines the benefits of self-monitoring and control of cholesterol levels for the first time.

The patients in the intervention arm will receive a device for self-measurement of cholesterol values and will be trained in its use. These patients will independently measure their cholesterol levels monthly using capillary blood tests and report the results to the study physicians, who will then adjust the therapy accordingly. The control arm is treated according to local standards, which includes control of the cholesterol values twice a year at the visit in out-patient clinic. Patients in both study arms will be followed up for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with acute coronary syndrome in the last 6 months and not having reached the LDL target value
* Signed informed consent

Exclusion Criteria:

* Persons unable to understand the study
* Persons unable or unwilling to perform self-measurements
* Persons unable or unwilling to undergo additional cholesterol-lowering therapy to reach the LDL target
* Pre-menopausal women without contraception
* Use of experimental drugs or investigational products within 30 days prior to screening
* Employees or contractors of the institution conducting the study or family members of the Principal Investigator, Co-Investigator, or financial supporter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
percentage value LDL-Cholesterol reduction in comparison to baseline | 6 months
  Compare the change in value of LDL-Cholesterol with additional monthly self measurement of parameters after 6 months versus baseline and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Laufs, Professor, Study Chair — University Clinik, Clinic for Cardiology Leipzig
Locations (1):
- Clinic of cardiology University clinic Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joseph P, Leong D, McKee M, Anand SS, Schwalm JD, Teo K, Mente A, Yusuf S. Reducing the Global Burden of Cardiovascular Disease, Part 1: The Epidemiology and Risk Factors. Circ Res. 2017 Sep 1;121(6):677-694. doi: 10.1161/CIRCRESAHA.117.308903. PMID 28860318
- [Background] Ference BA, Ginsberg HN, Graham I, Ray KK, Packard CJ, Bruckert E, Hegele RA, Krauss RM, Raal FJ, Schunkert H, Watts GF, Boren J, Fazio S, Horton JD, Masana L, Nicholls SJ, Nordestgaard BG, van de Sluis B, Taskinen MR, Tokgozoglu L, Landmesser U, Laufs U, Wiklund O, Stock JK, Chapman MJ, Catapano AL. Low-density lipoproteins cause atherosclerotic cardiovascular disease. 1. Evidence from genetic, epidemiologic, and clinical studies. A consensus statement from the European Atherosclerosis Society Consensus Panel. Eur Heart J. 2017 Aug 21;38(32):2459-2472. doi: 10.1093/eurheartj/ehx144. PMID 28444290
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Cholesterol Treatment Trialists' (CTT) Collaboration; Fulcher J, O'Connell R, Voysey M, Emberson J, Blackwell L, Mihaylova B, Simes J, Collins R, Kirby A, Colhoun H, Braunwald E, La Rosa J, Pedersen TR, Tonkin A, Davis B, Sleight P, Franzosi MG, Baigent C, Keech A. Efficacy and safety of LDL-lowering therapy among men and women: meta-analysis of individual data from 174,000 participants in 27 randomised trials. Lancet. 2015 Apr 11;385(9976):1397-405. doi: 10.1016/S0140-6736(14)61368-4. Epub 2015 Jan 9. PMID 25579834
- [Background] Cholesterol Treatment Trialists' (CTT) Collaborators; Mihaylova B, Emberson J, Blackwell L, Keech A, Simes J, Barnes EH, Voysey M, Gray A, Collins R, Baigent C. The effects of lowering LDL cholesterol with statin therapy in people at low risk of vascular disease: meta-analysis of individual data from 27 randomised trials. Lancet. 2012 Aug 11;380(9841):581-90. doi: 10.1016/S0140-6736(12)60367-5. Epub 2012 May 17. PMID 22607822
- [Background] Silverman MG, Ference BA, Im K, Wiviott SD, Giugliano RP, Grundy SM, Braunwald E, Sabatine MS. Association Between Lowering LDL-C and Cardiovascular Risk Reduction Among Different Therapeutic Interventions: A Systematic Review and Meta-analysis. JAMA. 2016 Sep 27;316(12):1289-97. doi: 10.1001/jama.2016.13985. PMID 27673306
- [Background] Kotseva K, De Backer G, De Bacquer D, Ryden L, Hoes A, Grobbee D, Maggioni A, Marques-Vidal P, Jennings C, Abreu A, Aguiar C, Badariene J, Bruthans J, Castro Conde A, Cifkova R, Crowley J, Davletov K, Deckers J, De Smedt D, De Sutter J, Dilic M, Dolzhenko M, Dzerve V, Erglis A, Fras Z, Gaita D, Gotcheva N, Heuschmann P, Hasan-Ali H, Jankowski P, Lalic N, Lehto S, Lovic D, Mancas S, Mellbin L, Milicic D, Mirrakhimov E, Oganov R, Pogosova N, Reiner Z, Stoerk S, Tokgozoglu L, Tsioufis C, Vulic D, Wood D; EUROASPIRE Investigators*. Lifestyle and impact on cardiovascular risk factor control in coronary patients across 27 countries: Results from the European Society of Cardiology ESC-EORP EUROASPIRE V registry. Eur J Prev Cardiol. 2019 May;26(8):824-835. doi: 10.1177/2047487318825350. Epub 2019 Feb 10. PMID 30739508
- [Background] Ray KK, Molemans B, Schoonen WM, Giovas P, Bray S, Kiru G, Murphy J, Banach M, De Servi S, Gaita D, Gouni-Berthold I, Hovingh GK, Jozwiak JJ, Jukema JW, Kiss RG, Kownator S, Iversen HK, Maher V, Masana L, Parkhomenko A, Peeters A, Clifford P, Raslova K, Siostrzonek P, Romeo S, Tousoulis D, Vlachopoulos C, Vrablik M, Catapano AL, Poulter NR; DA VINCI study. EU-Wide Cross-Sectional Observational Study of Lipid-Modifying Therapy Use in Secondary and Primary Care: the DA VINCI study. Eur J Prev Cardiol. 2021 Sep 20;28(11):1279-1289. doi: 10.1093/eurjpc/zwaa047. PMID 33580789
- [Background] Sturzebecher PE, Tunnemann-Tarr A, Tuppatsch K, Laufs U. [Treatment and LDL cholesterol adjustment in patients with high and very high cardiovascular risk in Germany compared with Europe - data from the SANTORINI registry]. Dtsch Med Wochenschr. 2023 Apr;148(9):55-64. doi: 10.1055/a-2009-5077. Epub 2023 Mar 1. German. PMID 36858065
- [Background] Fox KM, Tai MH, Kostev K, Hatz M, Qian Y, Laufs U. Treatment patterns and low-density lipoprotein cholesterol (LDL-C) goal attainment among patients receiving high- or moderate-intensity statins. Clin Res Cardiol. 2018 May;107(5):380-388. doi: 10.1007/s00392-017-1193-z. Epub 2017 Dec 22. PMID 29273856
- [Background] Cannon CP, Khan I, Klimchak AC, Reynolds MR, Sanchez RJ, Sasiela WJ. Simulation of Lipid-Lowering Therapy Intensification in a Population With Atherosclerotic Cardiovascular Disease. JAMA Cardiol. 2017 Sep 1;2(9):959-966. doi: 10.1001/jamacardio.2017.2289. PMID 28768335
- [Background] Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Z, Riccardi G, Taskinen MR, Tokgozoglu L, Verschuren WMM, Vlachopoulos C, Wood DA, Zamorano JL, Cooney MT; ESC Scientific Document Group. 2016 ESC/EAS Guidelines for the Management of Dyslipidaemias. Eur Heart J. 2016 Oct 14;37(39):2999-3058. doi: 10.1093/eurheartj/ehw272. Epub 2016 Aug 27. No abstract available. PMID 27567407
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Katzmann JL, Sorio-Vilela F, Dornstauder E, Fraas U, Smieszek T, Zappacosta S, Laufs U. Non-statin lipid-lowering therapy over time in very-high-risk patients: effectiveness of fixed-dose statin/ezetimibe compared to separate pill combination on LDL-C. Clin Res Cardiol. 2022 Mar;111(3):243-252. doi: 10.1007/s00392-020-01740-8. Epub 2020 Sep 19. PMID 32949286
- [Background] Alonso R, Cuevas A, Cafferata A. Diagnosis and Management of Statin Intolerance. J Atheroscler Thromb. 2019 Mar 1;26(3):207-215. doi: 10.5551/jat.RV17030. Epub 2019 Jan 19. PMID 30662020
- [Background] Jacobson TA. NLA Task Force on Statin Safety--2014 update. J Clin Lipidol. 2014 May-Jun;8(3 Suppl):S1-4. doi: 10.1016/j.jacl.2014.03.003. No abstract available. PMID 24793438
- [Background] Serban MC, Colantonio LD, Manthripragada AD, Monda KL, Bittner VA, Banach M, Chen L, Huang L, Dent R, Kent ST, Muntner P, Rosenson RS. Statin Intolerance and Risk of Coronary Heart Events and All-Cause Mortality Following Myocardial Infarction. J Am Coll Cardiol. 2017 Mar 21;69(11):1386-1395. doi: 10.1016/j.jacc.2016.12.036. PMID 28302290